CLINICAL TRIAL: NCT07009288
Title: Decreasing Cardiometabolic Risk in Childhood Cancer Survivors: The STRENGTH (Survivors Engaged in Time-Restricted EatiNG After THerapy) Study
Brief Title: A Study of Time-Restricted Eating in Childhood Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-250
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Childhood Cancer Survivors
MeSH Terms: interventions — Angptl4 protein, mouse; Dried Blood Spot Testing

STUDY DESIGN:
Intervention Model Description: This is a phase 2b randomized controlled trial of a TRE intervention among childhood cancer survivor participants with overweight and obesity in the Childhood Cancer Survivor Study (CCSS), designed according to the ORBIT model for behavioral intervention development.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Team members conducting data analysis will be blinded to each participant's assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will be instructed to participate in time-restricted eating, building to a 16-hour fast per day (not eating or drinking calorie-enriched beverages such as soda or nutritional shakes for a 16-hour window, such as 6pm -10am or 7pm-11am). These participants will also receive motivational phone/video calls with a trained health coach, daily text message reminders of when to start and stop their fasting, and monthly weight check-ins.
  Interventions: Other: Monthly weights; Other: Fasting; Other: Calls; Other: Participant Questionnaires; Other: Dried blood spot
- Control Group (Active Comparator): Participants will receive the standard of care electronic handouts through the Way to Health platform, and monthly weight check-ins.
  Interventions: Other: Children's Oncology Group Heart Health Link; Other: Monthly weights; Other: Dried blood spot

INTERVENTIONS:
Other: Children's Oncology Group Heart Health Link — Educational materials on healthy lifestyle behaviors.
  Arms: Control Group
Other: Monthly weights — Weight (kg): measured remotely via Withings Body + scale, Height, weight, waist circumference, BP, and % body fat
Other: Fasting — (14-hour fast x 2 weeks; 15-hour fast x- 1 week; 16-hour fast for the remainder of the active intervention)
  Arms: Intervention Group
Other: Calls — Month 1-3: Bi-weekly call using motivational interviewing Months 4-6: Monthly call using motivational interviewing Support via SMS text
  Arms: Intervention Group
Other: Participant Questionnaires — Questions on worry, perceived self-efficacy, health beliefs and knowledge of late effects (adapted from EQUAL study), Behavioral Risk Factor Surveillance System, Physical Activity Questionnaire, Link to Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool with accompanying sleep module
  Arms: Intervention Group
Other: Dried blood spot — Glucose, insulin, hemoglobin A1c, lipids. Measured remotely in the fasting state via dried blood spots in the participant's home.

SUMMARY:
This study will look at whether motivational sessions (including regular calls with a trained health coach) in combination with time-restricted eating (TRE) is an effective way to achieve weight loss and lower cardiometabolic risk in adult survivors of childhood cancer. The researchers will look at how effective this intervention is compared to the usual approach, which is to review educational materials and measure weight once a month. This study will not provide treatment for any disease or cancer.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Childhood Cancer Survivor Study (a cohort of 5+ year survivors of childhood cancer diagnosed at age < 21 between 1970-1999 at 31 participating institutions in North America)
* Are ≥18 years old
* Self-reported body mass index ≥ 25 kg/m2
* Are not pregnant or do not intend to become pregnant in the next year
* Stable weight over the past 3 months (+/- 10 pounds)
* If on oral medication for insulin resistance (ie, metformin), elevated blood pressure, or dyslipidemia, medication dose must be stable (ie, unchanged > 3 months)
* Have internet access (can be via smartphone or computer). If neither device is available, the study can loan participants a Wi-Fi enabled device.

Exclusion Criteria:

* Do not reside in the United States
* Do not speak English
* Already fasting >13 hours per 24-hour day
* On insulin or GLP-1 agonist
* Diagnosis of type 1 diabetes mellitus
* Enrolled in a formal weight management program or other weight loss trial
* History of an eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in weight | at 12 months

SECONDARY OUTCOMES:
Change in glucose | up to 12 months
  via dried blood spots
Change in insulin | up to 12 months
  via dried blood spots
Change in HbA1c | up to 12 months
  via dried blood spots

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Friedman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Hunter College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - St. Jude Children's Research Hospital (Data Collection Only), Memphis, Tennessee
  - Fred Hutchinson Cancer Research Center (Data Collection Only), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org